CLINICAL TRIAL: NCT06437769
Title: The Effect of Reiki Applied to Women Who Have Been Hospitalized by Cesarean During the Hospitalization Process on Anxiety, Depression, Comfort and Breastfeeding
Brief Title: The Effect of Reiki on Cesarean During Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/236
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): . Reiki therapy will be applied to the participants for 30 minutes while they lie down with their eyes closed. A total of 4 sessions of Reiki application will be applied to the intervention group at the 4th hour, 8th hour, 24th hour and 28th hour after the cesarean section. Reiki application will be applied at the 4th hour after the cesarean section. Comfort, anxiety, depression and breastfeeding symptoms after the 4th session will be recorded.
  Interventions: Other: reiki
- control group (No Intervention): will provided with standard midwifery care.

INTERVENTIONS:
Other: reiki — effect of reiki application to women who have been hospitalized by ceserean during the hospitlalization process on anxiety depression comfort and breastfeesing
  Other Names: control group
  Arms: Reiki

SUMMARY:
To determine the effect of reiki applied to women who have been hospitalized by cesarean during the hospitalization process on anxiety, depression, comfort and breastfeeding

Method: The study will be completed in a randomized controlled manner with a total of 70 women, 35 in the experimental group and 35 in the control group. Women in the experimental group Reiki therapy will be applied to the participants for 30 minutes while they lie down with their eyes closed. Research data will be collected with the Comfort Scale, Hospital anxiety and depression scale and bristol breastfeeding points and will be recorded

DETAILED DESCRIPTION:
Design and Settings: This randomized controlled experimental study will conducted in the post operative room of the, Turkey between the dates of June 2024 and October 2024

ELIGIBILITY:
Inclusion Criteria:

* volunteering
* be over 18 years old
* Not having a diagnosed psychiatric disease
* no communication problems
* No drug sensitivity or allergy
* women who have had a cesarean section

Exclusion Criteria:

* Having a diagnosed psychiatric illness
* no communication problems
* Being under 18 years of age
* not volunteering to participate in the research
* drug sensitivity and allergy
* women who gave birth normally

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
anxiety and depression | immediately after intervention
  Hospital Anxiety and Depression Scale;Hospital anxiety depression scale, to screen anxiety and depression in people with physical illnesses.
  has been prepared. It consists of 14 items.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye BAL, Ph.D., Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)